CLINICAL TRIAL: NCT05356949
Title: Effectiveness of Enhanced Mental Health Support for Young People
Acronym: Nopsatuki
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other); City of Turku (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12086-2020
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Depression; Anxiety; Emotional Stress
Keywords: Depression; Anxiety; Intervention; Adolescents; School
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress, Psychological | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The participants receive a psychological intervention including six weekly sessions. The intervention is based on methods of cognitive-behavioral therapy and delivered by a psychiatric nurse working in the participant's school.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — The participants receive a psychological intervention including six weekly sessions. The intervention is based on methods of cognitive-behavioral therapy and delivered by a psychiatric nurse working in the participant's school.

SUMMARY:
The aim of the research project is to measure the effectiveness of an early and rapid psychiatric nurse intervention at schools in improving the emotional well-being and functioning of adolescents.

DETAILED DESCRIPTION:
In this study, the impact of a short psychological intervention on adolescent emotional well-being, symptoms, and functioning is assessed. The intervention is a short intervention based on the methods of cognitive-behavioral therapy comprising 6 weekly sessions. It is delivered by psychiatric nurses working in the schools in the City of Turku. The participants are adolescents aged 12-18 who seek student health care due to mental health problems. The goal is to recruit 150 participants. The intervention is not tied to some particular disorder and thus, the main response variable is emotional well-being. Emotional well-being is measured at both the beginning and the end of the intervention, and at 6-month follow-up using the Young Person's Clinical Outcomes for Routine Evaluation (YP-CORE) questionnaire. Effectiveness is measured as a change in the YP-CORE scores.

ELIGIBILITY:
Inclusion Criteria:

* Young Person's Clinical Outcomes for Routine Evaluation (YP-CORE) score ≥14
* Willing and able to commit to the intervention and study protocol
* Sufficient proficiency in Finnish

Exclusion Criteria:

* Other ongoing mental health treatment
* Substance use as the main problem

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Emotional well-being, short-term | 6 weeks
  Change from the baseline to the end of the intervention in the Young Person's Clinical Outcomes for Routine Evaluation (YP-CORE) score. The score range for the scale is 0-40 and lower scores indicate better emotional well-being.

SECONDARY OUTCOMES:
Emotional well-being, long-term | 6 months
  Change from the baseline to the 6 month follow-up time-point in the Young Person's Clinical Outcomes for Routine Evaluation (YP-CORE) score. The score range for the scale is 0-40 and lower scores indicate better emotional well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Max Karukivi, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Southwest Finland, Finland

REFERENCES:
- [Derived] Tornivuori A, Kronstrom K, Aromaa M, Salantera S, Karukivi M. Accessible mental well-being intervention for adolescents in school settings: a single-group intervention study using a pretest-post-test design. Child Adolesc Psychiatry Ment Health. 2023 Feb 20;17(1):28. doi: 10.1186/s13034-023-00576-0. PMID 36805796